CLINICAL TRIAL: NCT04965922
Title: Quality of Life of Caregivers and Patients Suffering From Multiple System Atrophy
Acronym: QUA2-AMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2020/29
Record Dates: First submitted 2021-05-06; First posted 2021-07-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; Quality of life; Multimodal intervention; Neurodegenerative disease
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal intervention at inclusion (Experimental): Multimodal intervention will be proposed to Multiple system atrophy patients and their caregivers.
  Interventions: Behavioral: Multimodal intervention
- Multimodal intervention at 6 month (Other): Multimodal intervention will be proposed to Multiple system atrophy patients and their caregivers.
  Interventions: Behavioral: Multimodal intervention

INTERVENTIONS:
Behavioral: Multimodal intervention — The intervention consists of identifying the individual needs of each caregiver and patient and identifying sources of improvement in the management of daily life, including the optimization of social support. This optimization requires the involvement of people in the environment (family, friends, neighbours) who can provide help, support of any kind, recurrent or punctual, minimizing negative family interactions and maximizing positive contributions by each in supporting and supporting the individual.
  The intervention is personalized in the sense that the content of each session seeks to adapt itself to the specificities of the couple situation and its surroundings.
  interviews/meetings involving a psychologist social worker.

SUMMARY:
Multiple system atrophy (MSA) is a rare and fatal neurodegenerative disorder that cause as other neurodegenerative diseases profound declines in functioning and thus, require caregiving for assistance with daily living. The aim of the study is to evaluate the effect of a multimodal intervention as proposed by the NYU Caregiver Counseling and Support Intervention (NYUCI) on the quality of life of patients and their caregivers.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a rare and fatal neurodegenerative disorder, which is characterized by a variable combination of parkinsonism, cerebellar dysfunction, autonomic failure, and additional signs. No effective treatment is available. MSA patients have a poor prognosis with a median survival ranging between 6 and 10 years. MSA as other neurodegenerative diseases cause profound declines in functioning ; thus, many patients require caregivers for assistance with daily living. Caregiving can also be extremely stressful, and many caregivers experience declines in mental health. All of these repercussions contribute to the deterioration of the caregiver's quality of life and they can have an impact on the patient, in particular, on the patient's survival. Improving quality of life is a major element and identifying effective targeted interventions would bring immediate and direct benefit to patients and their families. In this context, it seems that a multimodal intervention as proposed by the NYU Caregiver Counseling and Support Intervention (NYUCI) developed by Mittelman could contribute to improve disease management and better coping with daily living difficulties. The NYUCI strategy combines sessions of individual and family counseling, support group participation, and additional on-call telephone consultations in a flexible counseling approach that is tailored to each caregiving family

ELIGIBILITY:
Patients Inclusion Criteria :

* Patients suffering from "possible" or "probable" MSA according to clinical consensus criteria
* Living at home
* Presence of at least one close person (family caregiver or not) in the entourage
* Unified Multiple System Atrophy Rating Scale (UMSARS) IV ≤4
* Written informed consent
* Patient covered by the national health system

Caregivers Inclusion Criteria :

* Age > 18
* Able to answer to study scales and survey
* Written informed consent

Patients Exclusion Criteria:

* Unified Multiple System Atrophy Rating Scale (UMSARS) IV > 4
* Absence of at least one close person

Caregivers Inclusion Criteria :

- Enable to answer to study scales and survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Multiple System Atrophy Quality of Life (MSA-QoL) Score | Day 0
  Score of emotional and social sub-dimension of the MSA Quality of Life scale. Quality of life questionnaire to collect the level of difficulty experienced by the patient (from no problem to extreme problem) during the 4 weeks preceding the interview on activities such as: moving; walking; maintaining balance; speak; feed oneself. It also assesses the patient's feelings about his illness.
Multiple System Atrophy Quality of Life (MSA-QoL) Score | 6 month
  Score of emotional and social sub-dimension of the MSA Quality of Life scale. Quality of life questionnaire to collect the level of difficulty experienced by the patient (from no problem to extreme problem) during the 4 weeks preceding the interview on activities such as: moving; walking; maintaining balance; speak; feed oneself. It also assesses the patient's feelings about his illness.
Multiple System Atrophy Quality of Life (MSA-QoL) Score | 12 month
  Score of emotional and social sub-dimension of the MSA Quality of Life scale. Quality of life questionnaire to collect the level of difficulty experienced by the patient (from no problem to extreme problem) during the 4 weeks preceding the interview on activities such as: moving; walking; maintaining balance; speak; feed oneself. It also assesses the patient's feelings about his illness.

SECONDARY OUTCOMES:
Center for Epidemiologic Sutdies-Depression (CESD) Score | Day 0
  20 items scale used to assess the existence of a depressive syndrome. Scores less than 15 does not indicate any depressive disorder Scores between 15 and 21 are indicative of mild to moderate depression. Scores above 21 are consistent with the existence of severe/ major depression
Center for Epidemiologic Sutdies-Depression (CESD) Score | 3 month
  20 items scale used to assess the existence of a depressive syndrome. Scores less than 15 does not indicate any depressive disorder Scores between 15 and 21 are indicative of mild to moderate depression. Scores above 21 are consistent with the existence of severe/ major depression
Center for Epidemiologic Sutdies-Depression (CESD) Score | 6 month
  20 items scale used to assess the existence of a depressive syndrome. Scores less than 15 does not indicate any depressive disorder Scores between 15 and 21 are indicative of mild to moderate depression. Scores above 21 are consistent with the existence of severe/ major depression
Multiple System Atrophy Quality of Life (MSA-QoL) Score | Day 0
  Score of other sub-dimension of the MSA Quality of Life scale. The MSA-QoL questionnaire is composed of three different subscales: motor (14 items), non-motor (12 items) and emotional/social (14 items). The response options for each question range from 0 (no problem) to 4 (extreme problem) with higher total scores reflecting more impaired quality of life. The MSA-QoL also includes a visual analogue scale (VAS) of how satisfied patients feel (range 0-100, with lower scores indicating lower quality of life).
Multiple System Atrophy Quality of Life (MSA-QoL) Score | 3 month
  Score of other sub-dimension of the MSA Quality of Life scale. The MSA-QoL questionnaire is composed of three different subscales: motor (14 items), non-motor (12 items) and emotional/social (14 items). The response options for each question range from 0 (no problem) to 4 (extreme problem) with higher total scores reflecting more impaired quality of life. The MSA-QoL also includes a visual analogue scale (VAS) of how satisfied patients feel (range 0-100, with lower scores indicating lower quality of life).
Multiple System Atrophy Quality of Life (MSA-QoL) Score | 6 month
  Score of other sub-dimension of the MSA Quality of Life scale. The MSA-QoL questionnaire is composed of three different subscales: motor (14 items), non-motor (12 items) and emotional/social (14 items). The response options for each question range from 0 (no problem) to 4 (extreme problem) with higher total scores reflecting more impaired quality of life. The MSA-QoL also includes a visual analogue scale (VAS) of how satisfied patients feel (range 0-100, with lower scores indicating lower quality of life).
State Trait Inventory Anxiety (STAI) Score | Day 0
  Anxiety assessment. 2 scales of 20 questions used to assess how subjects feel at the time and generally. Score > 65 means high anxiety ; Score < 35 means low anxiety
State Trait Inventory Anxiety (STAI) Score | 3 month
  Anxiety assessment. 2 scales of 20 questions used to assess how subjects feel at the time and generally. Score > 65 means high anxiety ; Score < 35 means low anxiety
State Trait Inventory Anxiety (STAI) Score | 6 month
  Anxiety assessment. 2 scales of 20 questions used to assess how subjects feel at the time and generally. Score > 65 means high anxiety ; Score < 35 means low anxiety
Unified Multiple System Atrophy Rating Scale (UMSARS) I | Day 0
  (0=no disorder, 48=severe disorders): Is an assessment of daily life activities via 12 12 items scale used to assess language, writing, autonomy , walking and the presence of possible urinary, sexual or intestinal disorders. (0=no disorder, 48=severe)
Unified Multiple System Atrophy Rating Scale (UMSARS) I | 3 month
  (0=no disorder, 48=severe disorders): Is an assessment of daily life activities via 12 12 items scale used to assess language, writing, autonomy , walking and the presence of possible urinary, sexual or intestinal disorders. (0=no disorder, 48=severe)
Unified Multiple System Atrophy Rating Scale (UMSARS) I | 6 month
  (0=no disorder, 48=severe disorders): Is an assessment of daily life activities via 12 12 items scale used to assess language, writing, autonomy , walking and the presence of possible urinary, sexual or intestinal disorders. (0=no disorder, 48=severe)
Unified Multiple System Atrophy Rating Scale (UMSARS) II | Day 0
  Motor examination based on 14 items that allow to evaluate in particular facial expression, oculomotricity, oral expression, tremors or walking. 0=no disorder, 56=severe disorders
Unified Multiple System Atrophy Rating Scale (UMSARS) II | 3 month
  Motor examination based on 14 items that allow to evaluate in particular facial expression, oculomotricity, oral expression, tremors or walking. 0=no disorder, 56=severe disorders
Unified Multiple System Atrophy Rating Scale (UMSARS) II | 6 month
  Motor examination based on 14 items that allow to evaluate in particular facial expression, oculomotricity, oral expression, tremors or walking. 0=no disorder, 56=severe disorders
Unified Multiple System Atrophy Rating Scale (UMSARS) III | Day 0
  Blood pressure and heart rate measurements in the lying and standing position for 10 min every minute.
Unified Multiple System Atrophy Rating Scale (UMSARS) III | 3 month
  Blood pressure and heart rate measurements in the lying and standing position for 10 min every minute.
Unified Multiple System Atrophy Rating Scale (UMSARS) III | 6 month
  Blood pressure and heart rate measurements in the lying and standing position for 10 min every minute.
Unified Multiple System Atrophy Rating Scale (UMSARS) IV | Day 0
  Assessment of the disability from 1 to 5. 1 = completely independent ; 5 = totally dependent
Unified Multiple System Atrophy Rating Scale (UMSARS) IV | 3 month
  Assessment of the disability from 1 to 5. 1 = completely independent ; 5 = totally dependent
Unified Multiple System Atrophy Rating Scale (UMSARS) IV | 6 month
  Assessment of the disability from 1 to 5. 1 = completely independent ; 5 = totally dependent
Montreal Cognitive Assessment (MoCA) Score | Day 0
  evaluates short-term memory, visuospatial skills, executive functions, attention, concentration, work memory, language, abstraction, computation, and time and space orientation. Cognitive impairment is assessed by the score on 30 points (27-30: no cognitive impairment; 21-26: mild).
Montreal Cognitive Assessment (MoCA) Score | 3 month
  evaluates short-term memory, visuospatial skills, executive functions, attention, concentration, work memory, language, abstraction, computation, and time and space orientation. Cognitive impairment is assessed by the score on 30 points (27-30: no cognitive impairment; 21-26: mild).
Montreal Cognitive Assessment (MoCA) Score | 6 month
  evaluates short-term memory, visuospatial skills, executive functions, attention, concentration, work memory, language, abstraction, computation, and time and space orientation. Cognitive impairment is assessed by the score on 30 points (27-30: no cognitive impairment; 21-26: mild).
Zarit Scale score | Day 0
  Assesses caregiver burden. 22 item scale with total score ranging from 0 to 88. Score 20 mean zero load - Score > 60 means severe load
Zarit Scale score | 3 month
  Assesses caregiver burden. 22 item scale with total score ranging from 0 to 88. Score 20 mean zero load - Score > 60 means severe load
Zarit Scale score | 6 month
  Assesses caregiver burden. 22 item scale with total score ranging from 0 to 88. Score 20 mean zero load - Score > 60 means severe load
Family Relations Index (FRI) | Day 0
  27 items used to assess family functioning : family cohesion, verbalization of feelings and family conflict.
Family Relations Index (FRI) | 3 month
  27 items used to assess family functioning : family cohesion, verbalization of feelings and family conflict.
Family Relations Index (FRI) | 6 month
  27 items used to assess family functioning : family cohesion, verbalization of feelings and family conflict.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra FOUBERT-SAMIER, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux, Bordeaux, France